CLINICAL TRIAL: NCT03726086
Title: Post-extubation Assessment of Laryngeal Symptoms and Severity
Acronym: PALSS
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00151643; R01NR017433-01A1 (NIH)
Record Dates: First submitted 2018-10-26; First posted 2018-10-31 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Intubation, Intratracheal; Critical Illness; Mechanical Ventilation Complication; Complication of Ventilation Therapy
Keywords: larynx; injury; voice; trachea
MeSH Terms: conditions — Critical Illness; Laryngeal Diseases; Wounds and Injuries; Tracheal Diseases | interventions — Laryngoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: laryngoscopy — A flexible camera (fiberoptic endoscope) is placed in the patient's nose to view the nose, throat, and airway.

SUMMARY:
The goal of this study is to learn more about voice and airway problems that patients experience during and after the time patients have an oral endotracheal tube in patients' airway to help patients breathe while receiving mechanical ventilation in an intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Required mechanical ventilation via an oral endotracheal tube
* Anticipated intubation ≥8 hours

Exclusion Criteria:

* Pre-existing dysphonia, dysphagia
* Pre-existing central nervous system, neuromuscular, or connective tissue disease
* Prior tracheotomy and/or tracheotomy placed prior to enrollment
* History of major thoracic surgery (e.g., sternotomy, thoracotomy) prior to the current admission
* Head and/or neck disease
* Head and/or neck surgery other than tonsillectomy
* Known or suspected anatomical abnormalities or pre-intubation trauma of the oral cavity, pharynx, larynx, or esophagus
* Unlikely to be extubated (i.e., expected death)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit (ICU) who are orally intubated with mechanical ventilaton meeting inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Laryngeal injury as assessed by 4-point categorical scale | Within 72 hours post-extubation
  Characterize injuries to the larynx and surrounding tissues/anatomy after mechanical ventilation is no longer required and the oral endotracheal tube is removed. Injuries will be graded on a 4-point categorical scale ranging from 0 (no injury) to 3 (severe injury).
Laryngeal injury symptom grading by Laryngeal Hypersensitivity Questionnaire (LHQ) | Within 48 hours of anticipated extubation
  Characterize patient symptoms of laryngeal injury within 48 hours of anticipated extubation. Symptoms will be assessed using a 4-point ordinal scale based on the LHQ, ranging from 1 (all of the time) to 4 (none of the time).
Laryngeal injury symptom grading by LHQ | Within 72 hours post-extubation
  Characterize patient symptoms of laryngeal injury within 72 hours post-extubation. Symptoms will be assessed using a 4-point ordinal scale based on the LHQ, ranging from 1 (all of the time) to 4 (none of the time).
Laryngeal injury symptom grading by LHQ | 7 days post-extubation or hospital discharge, whichever occurs first
  Characterize patient symptoms of laryngeal injury at 7 days post-extubation or at discharge whichever comes first. Symptoms will be assessed using a 4-point ordinal scale based on the LHQ, ranging from 1 (all of the time) to 4 (none of the time).

SECONDARY OUTCOMES:
Oral endotracheal tube size | At the time of intubation (directly following study enrollment)
  Size of the endotracheal tube
Duration of orotracheal intubation | From date of intubation to date of extubation or placement of a tracheostomy tube, whichever occurs first, assessed up to 14 days
  Number of days from placement to extubation of the oral endotracheal tube
Perceptual voice characteristics as assessed by Grade Rough Breathy Asthenic Strained (GRBAS) method | Within 72 hours post-extubation
  Assessed from standardized voice samples and digital recordings using the grade, rough, breathy, asthenic, and strained (GRBAS) method with a 4-point ordinal scale ranging from 0 (normal) to 3 (severe).
Perceptual voice characteristics as assessed by GRBAS method | 7 days post-extubation or hospital discharge, whichever occurs first
  Assessed from standardized voice samples and digital recordings using the grade, rough, breathy, asthenic, and strained (GRBAS) method with a 4-point ordinal scale ranging from 0 (normal) to 3 (severe).
Acoustic voice measurement as assessed by voice analysis software | Within 72 hours post-extubation
  Assessed from standardized voice samples and digital recordings using the Computerized Speech Lab (PENTAX Medical) with voice analysis software (viz., Multi-Dimensional Voice Program (MDVP); Analysis of Dysphonia in Speech and Voice (ADSV)) to quantify voice characteristics across a number of parameters
Acoustic voice measurement as assessed by voice analysis software | 7 days post-extubation or hospital discharge, whichever occurs first
  Assessed from standardized voice samples and digital recordings using the Computerized Speech Lab (PENTAX Medical) with voice analysis software (viz., Multi-Dimensional Voice Program (MDVP); Analysis of Dysphonia in Speech and Voice (ADSV)) to quantify voice characteristics across a number of parameters.
Patient perception of voice and voice symptoms assessed by the Voice Symptom Scale (VoiSS) | Within 72 hours post-extubation and at 7 days post-extubation or hospital discharge, whichever occurs first
  a 30-item questionnaire that uses scaled scores across 3 domains-impairment (15 items), physical symptoms (8 items), and emotional response (7 items).
Isometric Hand Grip Strength-Dynamometry | Within 48 hours of anticipated extubation, within 72 hours post-extubation, and at 7 days post-extubation or hospital discharge, whichever occurs first
  Grip strength provides a measure of distal muscle strength that has important functional application for patients. Grip strength, tested by hand grip dynamometry, will be assessed in each hand using a Jamar Preston hand dynamometer
Peak tongue strength assessed using the Iowa Oral Performance Instrument (IOPI) | Within 48 hours of anticipated extubation, within 72 hours post-extubation, and at 7 days post-extubation or hospital discharge, whichever occurs first
  Tongue strength, tested using tongue bulb pressure, will be assessed using the Iowa Oral Performance Instrument (IOPI)
Yale Swallow Protocol | Within 72 hours post-extubation
  A cognitive screen and administration of a cup containing 3 oz. (90 ml) of water handed to the patient for uninterrupted continuous consumption via cup or straw. Interrupted consumption (i.e., stopping, resting), and/or coughing, choking, throat clearing, or a change in vocal quality (i.e., a wet, gurgly quality after consumption is completed) signifies a failed screening.
Function Oral Intake Scale (FOIS) | Within 90 days of extubation or at ICU discharge, whichever occurs first
  A 7-point clinical scale to document change in functional oral intake of food and liquid in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dale M. Needham, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adhikari NK, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. Lancet. 2010 Oct 16;376(9749):1339-46. doi: 10.1016/S0140-6736(10)60446-1. Epub 2010 Oct 11. PMID 20934212
- [Background] Balas MC, Vasilevskis EE, Burke WJ, Boehm L, Pun BT, Olsen KM, Peitz GJ, Ely EW. Critical care nurses' role in implementing the "ABCDE bundle" into practice. Crit Care Nurse. 2012 Apr;32(2):35-8, 40-7; quiz 48. doi: 10.4037/ccn2012229. PMID 22467611
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Benjamin B. Prolonged intubation injuries of the larynx: endoscopic diagnosis, classification, and treatment. Ann Otol Rhinol Laryngol Suppl. 1993 Apr;160:1-15. doi: 10.1177/00034894931020s401. PMID 8470867
- [Background] Bishop MJ, Weymuller EA Jr, Fink BR. Laryngeal effects of prolonged intubation. Anesth Analg. 1984 Mar;63(3):335-42. No abstract available. PMID 6367543
- [Background] Brandwein M, Abramson AL, Shikowitz MJ. Bilateral vocal cord paralysis following endotracheal intubation. Arch Otolaryngol Head Neck Surg. 1986 Aug;112(8):877-82. doi: 10.1001/archotol.1986.03780080077018. PMID 3718696
- [Background] Brodsky MB, Levy MJ, Jedlanek E, Pandian V, Blackford B, Price C, Cole G, Hillel AT, Best SR, Akst LM. Laryngeal Injury and Upper Airway Symptoms After Oral Endotracheal Intubation With Mechanical Ventilation During Critical Care: A Systematic Review. Crit Care Med. 2018 Dec;46(12):2010-2017. doi: 10.1097/CCM.0000000000003368. PMID 30096101
- [Background] Colice GL, Stukel TA, Dain B. Laryngeal complications of prolonged intubation. Chest. 1989 Oct;96(4):877-84. doi: 10.1378/chest.96.4.877. PMID 2791687
- [Background] Colice GL. Resolution of laryngeal injury following translaryngeal intubation. Am Rev Respir Dis. 1992 Feb;145(2 Pt 1):361-4. doi: 10.1164/ajrccm/145.2_Pt_1.361. PMID 1736742
- [Background] Donnelly WH. Histopathology of endotracheal intubation. An autopsy study of 99 cases. Arch Pathol. 1969 Nov;88(5):511-20. No abstract available. PMID 5347141
- [Background] Dubick MN, Wright BD. Comparison of laryngeal pathology following long-term oral and nasal endotracheal intubations. Anesth Analg. 1978 Nov-Dec;57(6):663-8. No abstract available. PMID 569990
- [Background] Eckerbom B, Lindholm CE, Alexopoulos C. Airway lesions caused by prolonged intubation with standard and with anatomically shaped tracheal tubes. A post-mortem study. Acta Anaesthesiol Scand. 1986 Jul;30(5):366-73. doi: 10.1111/j.1399-6576.1986.tb02432.x. PMID 3766091
- [Background] Hamdan AL, Sabra O, Rameh C, El-Khatib M. Persistant dysphonia following endotracheal intubation. Middle East J Anaesthesiol. 2007 Feb;19(1):5-13. PMID 17511179
- [Background] Hamdan AL, Sibai A, Rameh C, Kanazeh G. Short-term effects of endotracheal intubation on voice. J Voice. 2007 Nov;21(6):762-8. doi: 10.1016/j.jvoice.2006.06.003. Epub 2006 Aug 14. PMID 16905292
- [Background] Massard G, Rouge C, Dabbagh A, Kessler R, Hentz JG, Roeslin N, Wihlm JM, Morand G. Tracheobronchial lacerations after intubation and tracheostomy. Ann Thorac Surg. 1996 May;61(5):1483-7. doi: 10.1016/0003-4975(96)00083-5. PMID 8633963
- [Background] Pandian V, Thompson CB, Feller-Kopman DJ, Mirski MA. Development and validation of a quality-of-life questionnaire for mechanically ventilated ICU patients. Crit Care Med. 2015 Jan;43(1):142-8. doi: 10.1097/CCM.0000000000000552. PMID 25072754
- [Background] Sadoughi B, Fried MP, Sulica L, Blitzer A. Hoarseness evaluation: a transatlantic survey of laryngeal experts. Laryngoscope. 2014 Jan;124(1):221-6. doi: 10.1002/lary.24178. Epub 2013 Jun 26. PMID 23804513
- [Background] Santos PM, Afrassiabi A, Weymuller EA Jr. Prospective studies evaluating the standard endotracheal tube and a prototype endotracheal tube. Ann Otol Rhinol Laryngol. 1989 Dec;98(12 Pt 1):935-40. doi: 10.1177/000348948909801204. PMID 2589761
- [Background] Santos PM, Afrassiabi A, Weymuller EA Jr. Risk factors associated with prolonged intubation and laryngeal injury. Otolaryngol Head Neck Surg. 1994 Oct;111(4):453-9. doi: 10.1177/019459989411100411. PMID 7936678
- [Background] Scheel R, Pisegna JM, McNally E, Noordzij JP, Langmore SE. Endoscopic Assessment of Swallowing After Prolonged Intubation in the ICU Setting. Ann Otol Rhinol Laryngol. 2016 Jan;125(1):43-52. doi: 10.1177/0003489415596755. Epub 2015 Jul 26. PMID 26215724
- [Background] Tadie JM, Behm E, Lecuyer L, Benhmamed R, Hans S, Brasnu D, Diehl JL, Fagon JY, Guerot E. Post-intubation laryngeal injuries and extubation failure: a fiberoptic endoscopic study. Intensive Care Med. 2010 Jun;36(6):991-8. doi: 10.1007/s00134-010-1847-z. Epub 2010 Mar 18. PMID 20237758
- [Background] Tate JA, Sereika S, Divirgilio D, Nilsen M, Demerci J, Campbell G, Happ MB. Symptom communication during critical illness: the impact of age, delirium, and delirium presentation. J Gerontol Nurs. 2013 Aug;39(8):28-38. doi: 10.3928/00989134-20130530-03. Epub 2013 Jun 10. PMID 23755732